CLINICAL TRIAL: NCT06582849
Title: Enhanced Assistance During Radiotherapy for Unmet Essential Needs (EARN): a Single Center Hybrid Type 1 Efficacy-implementation Study
Brief Title: Enhanced Assistance During Radiotherapy for Unmet Essential Needs
Acronym: EARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202408150
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Bone Cancer; Brain Cancer; Colorectal Cancer; Esophagus Cancer; Lymphoma; Salivary Gland Cancer; Head and Neck Cancer; Liver Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Small Intestine Cancer; Stomach Cancer; Urinary Bladder Cancer; Anal Cancer; Blood Cancer; Breast Cancer; Cervical Cancer; Lung Cancer; Kidney Cancer; Penile Cancer; Skin Cancer; Testicular Cancer; Thyroid Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: Financial assistance; Health-related social needs; Social determinants of health; Radiotherapy; Cancer
MeSH Terms: conditions — Bone Neoplasms; Brain Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Lymphoma; Salivary Gland Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Urinary Bladder Neoplasms; Anus Neoplasms; Hematologic Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms; Kidney Neoplasms; Penile Neoplasms; Skin Neoplasms; Testicular Neoplasms; Thyroid Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard Assistance + Enhanced Assistance (Experimental): In the time period that patients are receiving radiotherapy, study participants will receive standard plus enhanced financial assistance for unmet essential needs.
  Interventions: Other: Standard assistance; Other: Enhanced assistance

INTERVENTIONS:
Other: Standard assistance — Standard assistance includes all community and institutional resources currently available for which the participant qualifies.
Other: Enhanced assistance — Enhanced assistance includes gift cards and checks to support food, housing, utilities, transportation, pharmacy, and other non-medical costs

SUMMARY:
This is a prospective single-arm study of an enhanced assistance intervention for patients with unmet essential needs undergoing >10 fractions of radiotherapy comparing delay-free completion of radiotherapy in study participants to historic controls.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Planned to receive or currently receiving a protracted course of curative-intent (neoadjuvant, definitive, or postoperative) radiotherapy.

  * For the purposes of this study, radiotherapy must consist of >10 fractions (if radiotherapy not yet initiated) or >15 additional fractions after the date of consent (if radiotherapy initiated prior to study consent).
* Be willing to undergo radiotherapy at the Barnes-Jewish Hospital location.
* Indicate at least 1 unmet essential need, including food insecurity, transportation insecurity, housing instability, utility needs, childcare needs, or other financial insecurity.
* Accept a referral to and meet with a social worker.
* Have unmet essential needs that will not be able to be fully addressed by standard assistance. This determination can be made by the assigned social worker or by the patient after they meet with the social worker.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Planned or scheduled to undergo radiotherapy simulation more than 28 days from the date of consent.
* Admitted to the hospital and not expected to undergo >10 fractions of radiotherapy as an outpatient.
* Undergoing treatment for anaplastic thyroid cancer. Patients with anaplastic thyroid cancer have a relatively low likelihood of completing radiotherapy due to the aggressive disease course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Delay-free completion of radiotherapy | Through completion of radiotherapy (estimated to be 4 months)
  Defined as: (1) completing all fractions of radiotherapy AND (2) delaying fewer than 5 fractions. Patients who do not initiate a recommended course of radiotherapy will be considered as not completing radiotherapy; however, in the rare case where the patient's radiotherapy treatment recommendation changes by their physician(s) to no longer include radiotherapy, such patients will be dropped from the study and excluded from analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Yang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu